CLINICAL TRIAL: NCT00163631
Title: Relationship of Vasoactive Peptide Levels to Portal Pressure and Patient Outcomes in Patients With Hepatic Cirrhosis
Status: Completed | Type: Observational
Sponsor: Bayside Health (Other Government)
Other Study IDs: 4104
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2006-10-04 (Estimated); Status verified 2005-09

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Investigate vasoactive medicators in portal hypertension on stored sera

ELIGIBILITY:
Inclusion Criteria:

* portal hypertension

Exclusion Criteria:

* Nil

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: William W Kemp, MBBS FRACP, Principal Investigator — The Alfred
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia